CLINICAL TRIAL: NCT03988972
Title: Efficacy of Diathermy on Healing Power of Cesarean Section Scar:A Randomized Control Trail
Brief Title: Efficacy of Diathermy on Healing Power of Cesarean Section Scar
Acronym: EDHPCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed abd elfatah elsenity, Lecturer of obstetrics and gynecology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 27180413
Record Dates: First submitted 2019-06-11; First posted 2019-06-18 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Healing Surgical Wounds
MeSH Terms: interventions — Diathermy; Laser Therapy

STUDY DESIGN:
Intervention Model Description: The 180 patients who will be included in our study will be randomized through computer generated system in to 2 groups. Group D (diathermy) and group S (scalpel). Each group will include 90 patients.
  Allocation and concealment will be done by sequentially sealed opaque envelopes. 180 envelopes will be numbered serially from 1 to 180, 90 envelopes will contain the letter D and the other 90 will contain the letter S.
  In each envelope, the corresponding letter which donates the allocated group will be put according to the randomization table and them all envelopes will be closed and put in one box. When the first patient arrives, the first envelope will be opened and the patient will be allocated according to the letter inside, whom will be allocated by a person not involved in the study.
Who Masked: Care Provider, Investigator
Masking Description: allocation done by a person not involved in the study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- diathermy group (Experimental): Diathermy incisions will be carried out using monopolar blade pen electrode, set on cutting mode and delivering a 35 continuous current. Electrosurgical cutting was performed without pressure or mechanical displacement.
  'Bleeders' will be controlled by using diathermy, on coagulating mode, and will be applied to a hemostat on the vessels
  Interventions: Device: diathermy
- scalpel group (Active Comparator): Incisions made by the scalpel will be done by the traditional method, with proper hemostasis by application of pressure to skin blood vessels and by ligating the subcutaneous bleeders.
  Interventions: Device: scalpel

INTERVENTIONS:
Device: diathermy — In women undergoing C.S, is healing power after diathermy equally to healing power after scalpel?
  Other Names: electro-cautrey
  Arms: diathermy group
Device: scalpel — Incisions made by the scalpel will be done by the traditional method, with proper hemostasis by application of pressure to skin blood vessels and by ligating the subcutaneous bleeders.
  Arms: scalpel group

SUMMARY:
To compare the effects of electro-surgery on healing power as a primary outcome (from skin to the peritoneum. And volume of blood loss, incision time and postoperative surgical wound pain as secondary outcomes.

DETAILED DESCRIPTION:
This is a prospective study is carried out at Ain Shams University Maternity Hospital, Obstetrics and Gynecology Department, Faculty of medicine in women undergoing CS through pfannentiel incisions.

All women will receive intravenous antibiotic prophylaxis according to the Ain Shams guideline, 1 g of cefazolin given at the time of incision.

Diathermy incisions will be carried out using monopolar blade pen electrode, set on cutting mode and delivering a 35 continuous current. Electrosurgical cutting will be performed without pressure or mechanical displacement.

'Bleeders' will be controlled by using diathermy, on coagulating mode, and will be applied to a hemostat on the vessels.

Incisions made by the scalpel will be done by the traditional method, with proper hemostasis by application of pressure to skin blood vessels and by ligating the subcutaneous bleeders.

After the operation and during the postoperative period, paracetamol (10mg/mL) 50-mL vial will be administered by i.v. infusion for analgesia on demand according to the patient's need with a 500-mg dose. And the wound will be sutured subcuticle by a prolene 3.0 sutures.

ELIGIBILITY:
Inclusion Criteria:

* Primi-section
* BMI (18-29) kg/m^2.
* Age from (18-40).
* Women undergoing CS with Pfannenstiel incision.

Exclusion Criteria:

* Women with one of the following conditions:

Patients requiring midline incision or on anti-coagulant therapy

* Cardiac patients on pacemakers and patients with chronic diseases expected to affect wound healing, such as diabetes, liver diseases, chronic anemia and renal impairment
* Obese patients BMI (>30) kg/m^2.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Cosmosis | 15 days after CS
  The primary objective is to compare healing power between two methods then will be followed at 3, 7, 11, and 15 days post-operative using: Visual Analogue Scale The original VAS consisted of a 100-mm line with "worst scar" at the right end of the line and "best scar" at the left end of the line. In this study, VAS ranged from 0 to 10cm. Using the line as a continuous entity, the patient mark on the line where they thought the scar fit.
Healing power | 15 days after cs
  The wound score addresses 6 clinical variables: absence of stepoff, contour ir- regularities, wound margin separation >2 mm, edge inversion, excessive distortion, and overall cosmetic appearance. Each of these categories is graded on a O-or-l-point scale. A total cosmetic score is derived by the addition of the scores of the 6 categorical variables. A score of 6 is considered optimal, while a score of ≤5 suboptimal.

SECONDARY OUTCOMES:
postoperative surgical wound pain: VAS scale | 24 hours
  postoperative surgical wound pain using visual analogue scale (VAS) after 1, 4,6,12 and 24 hours postoperatively. The visual analogue pain scale is a uni-dimensional measure of pain intensity, which has been used in adults. The visual analogue pain scale is an easy assessment tool consisting of a 10 cm line with 0 on one end, representing no pain, and 10 on the other end, representing the worst pain felt.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed abd elfatah elsenity, lecturer, Principal Investigator — Ain Shams University
Locations (1):
- Ain shams maternity teaching hospital, Cairo, Abbasia, Egypt

IPD SHARING:
Plan to Share IPD: No
will be shared in amaster sheet